CLINICAL TRIAL: NCT03678779
Title: Snack It Up for Parents: Interventions to Improve Children's Snacks
Acronym: SIU4P
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: Newman's Own Foundation (Unknown); Stop & Shop Supermarket Company (Unknown); Soccer4Success/America SCORES (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1601028
Record Dates: First submitted 2018-07-23; First posted 2018-09-20 (Actual); Last update posted 2018-09-20 (Actual); Status verified 2018-09

CONDITIONS: Snacking
Keywords: child nutrition; nutrition education; parent intervention
MeSH Terms: interventions — Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Incentive (Experimental): Each week parents received one $5 grocery store gift card per child in the household, intended for the purchase of healthy snacks, donated to the study by a partnering grocery store
  Interventions: Behavioral: Incentive
- Education (Experimental): Parents received brief weekly nutrition education videos (approximately one minute in length, uploaded on YouTube and viewable on most operating systems and on mobile devices
  Interventions: Behavioral: Education
- Combined (Experimental): Parents received both the Incentive and Education arm interventions
  Interventions: Behavioral: Combined

INTERVENTIONS:
Behavioral: Incentive — $5 grocery gift card
  Arms: Incentive
Behavioral: Education — Video-based brief nutrition education
  Arms: Education
Behavioral: Combined — Both Incentive and Education interventions received
  Arms: Combined

SUMMARY:
Influencing children's snacking habits has the potential to reap long-term rewards, yet few studies have focused on helping parents to provide healthier snacks for their children. The study tested the feasibility and preliminary effectiveness of parent interventions to improve snacks for children ages 8-12.

DETAILED DESCRIPTION:
Objective. Influencing children's snacking habits has the potential to reap long-term rewards, yet few studies have focused on helping parents to provide healthier snacks for their children. The study tested the feasibility and preliminary effectiveness of parent interventions to improve snacks for children ages 8-12.

Methods. Parents of children enrolled in an out-of-school-time soccer program in a low-income school district (n 16) were recruited. A comparison of 3 randomly-assigned interventions was conducted: 4 parents received grocery store gift cards (Incentive); 7 received nutrition education videos with tip sheets (Education); and 5 received both (Combined). The interventions were assessed qualitatively by interviewing parents and quantitatively to determine motivation (psychosocial survey) and children's snack quality (web-based 24-hour recall).

ELIGIBILITY:
Inclusion Criteria:

* 18 year and older
* Must have a child enrolled in one of three designated soccer sites of the study and must agree to let their child take the online 24 hour recall (ASA24)
* Must have a child 7 years or older participating on a soccer team
* Must frequently buy groceries from Stop & Shop (only if recruited for a study arms that involves grocery coupons)
* Must be literate in English or Spanish.

Exclusion Criteria:

* Failure to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-03 (Actual); Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
snack quality by on-line 24-hour dietary recall (ASA24) | 6 weeks
  grams of sugar, fruits and vegetables as snacks

SECONDARY OUTCOMES:
Intrinsic motivation by adapted Intrinsic Motivation Inventory | 6 weeks
  Parent intrinsic motivation for providing fruit and vegetable snacks; questions adapted from the Intrinsic Motivation Inventory (McAuley, E., Duncan, T., & Tammen, V. (1989). Psychometric properties of the Intrinsic Motivation Inventory in a competitive sport setting: A confirmatory factor analysis. Research Quarterly for Exercise and Sport, 60(1), 48-58).
Decisional balance by the Mainvil Decisional Balance Scale | 6 weeks
  Parent pros and cons for providing fruit and vegetable snacks to children; questions adapted from Mainvil decisional balance scale (Mainvil, L. A., Lawson, R., Horwath, C. C., McKenzie, J. E., & Hart, I. (2010). Validated scales to assess adult decisional balance to eat more fruits and vegetables. Appetite, 55(3), 454-465. doi:10.1016/j.appet.2010.08.007)
Self-efficacy by questions adapted NCI Food Attitudes and Behaviors Survey | 6 weeks
  Parent self-efficacy for providing fruit and vegetable snacks; questions adapted from the self-efficacy questions in the National Cancer Institute's Food Attitudes and Behaviors Survey (Erinosho, T. O., Pinard, C. A., Nebeling, L. C., Moser, R. P., Shaikh, A. R., Resnicow, K., . . . Yaroch, A. L. (2015). Development and implementation of the National Cancer Institute's Food Attitudes and Behaviors Survey to assess correlates of fruit and vegetable intake in adults. PLoS One, 10(2), e0115017. doi:10.1371/journal.pone.0115017)

IPD SHARING:
Plan to Share IPD: No